CLINICAL TRIAL: NCT01852760
Title: Assessment of Disease Activity in Ulcerative Colitis by Endoscopic Ultrasound
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other); University of Calgary (Other); University of Toronto (Other); Dalhousie University (Other)
Responsible Party: Principal Investigator, Brian Yan, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: UWO103563
Record Dates: First submitted 2013-05-07; First posted 2013-05-14 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Disease
Keywords: endoscopic ultrasound; ulcerative colitis; inflammatory bowel disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- UC in Remission: Patients with UC in remission
- UC Mild Disease: Patients with mild UC disease activity based on partial Mayo Score
- UC Moderate to severe: Patients with ulcerative colitis with moderate to severe disease activity based on partial Mayo score

SUMMARY:
In this cross-sectional study patients with active or quiescent ulcerative colitis will be studied to determine the utility of endoscopic ultrasound measurements of rectal wall blood flow and thickness as reliable indices of disease severity and the degree of correlation that exists with validated clinical, endoscopic, and histological indices.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a chronic inflammatory bowel disease (IBD) of unknown etiology characterized by diffuse mucosal inflammation limited to the colon. The basis of medical treatment is with agents that reduce the inflammatory process. Tailoring appropriate therapy will depend on disease severity, which can be difficult to identify. A response to therapy may also require months to determine. Medications for induction of remission and/or for maintenance in patients with mild to severe UC include 5-aminosalicylates (5'ASA), corticosteroids, azathioprine (AZA), cyclosporine, and infliximab (IFX). All medications have their own inherent side effect profile. Cost can be a major issue with some medications such as IFX, which can be tens of thousands of dollars annually. Medical management can still fail in those with severe disease necessitating surgical management with a colectomy. Identification of high-risk patients who are candidates for more intensive therapy early in the disease course might be a strategy to improve treatment outcomes and limit cost.

This notion of "individualizing" therapy is attractive and a distinct departure from the current "step-care" paradigm in which treatments are added sequentially on the basis of symptom-defined treatment failure. However, for this paradigm to be implementable an objective means of accurately stratifying risk must be identified and validated. Accordingly, increased interest has evolved in the use of biomarkers as prognostic tools. Although fecal calprotectin and serum CRP are potential candidates for this role, these tests have limitations.

Transabdominal ultrasound (US) has been used in the diagnostic workup of IBD. US was a good surrogate of disease activity when compared to colonoscopy, but is unable to reliably assess the rectal wall which tends to cause the most symptoms in UC. Endoscopic ultrasound (EUS) is a highly accurate diagnostic modality for the assessment of rectal pathology. However, the role of EUS in IBD is not well defined. Tsuga et al showed total wall thickness to be highly predictive for acute inflammation in patients with UC compared to healthy controls and that the degree of rectal wall involvement correlated with endoscopic severity. Higaki et al showed patients with quiescent UC who relapsed had initial sonographic evidence of "deep" disease activity shown by significantly greater baseline thickness of the first 3 layers of the rectal wall. Yoshizawa et al subsequently demonstrated that inflammation reaching the muscularis propria or deeper predicted the need for colectomy. Hurlstone et al correlated EUS scores with histopathology, endoscopic, and clinical scores and found good concordance to only exist with superficial EUS scores. In all of these studies the investigators who performed the EUS analysis did so with knowledge of the endoscopy scores. This questions the validity of these results due to the potential for bias. Another parameter that shows promise for evaluation of inflammatory burden is EUS evaluation of blood flow. Surprisingly, Doppler flow has not been used to assess bowel wall vascularity in UC with EUS. We believe that assessment of vascularity has the potential to differentiate with a high degree of accuracy active from quiescent disease.

Although the existing literature indicates that EUS has potential as an evaluative and prognostic tool the investigators believe that a great deal of additional research is needed to further develop this technology. This study will correlate Doppler EUS and other EUS indices with validated clinical, endoscopic, and histological indices of UC inflammation to assess its utility as a diagnostic tool. It will assess the reproducibility of these indices by calculating inter and intra-observer agreement by blinded expert reviewers. This information may have prognostic importance and might ultimately be used to guide therapy in individual patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of ulcerative colitis aged 18-85
* Patients termed either "active" or "inactive" UC
* Patients may be treatment naïve (ie: new diagnosis) or on existing therapy including 5'ASA (oral or topical), AZA, corticosteroids, or IFX

Exclusion Criteria:

* Inability to or unwillingness to undergo flexible sigmoidoscopy or colonoscopy
* Inability to provide informed consent
* Crohn's disease 4. Presence of an ileoanal pouch

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients with IBD attending outpatient IBD clinics at the University of Western Ontario teaching hospitals and patients admitted to hospital with severe UC will be included for endoscopic ultrasound assessment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The correlation between EUS indices, clinical, endoscopic, and histological scores of inflammation in UC | 1 day
  The correlation between EUS indices, clinical, endoscopic, and histological scores of inflammation in UC

SECONDARY OUTCOMES:
Interobserver variability of endoscopic and histologic scores | 1 day
  The agreement by raters of endoscopic and histologic scores of inflammation in UC using the intra-rater and inter-rater reliability.
Interobserver variability of EUS Indices | 1 day
  The agreement by rater's of EUS indices of inflammation using the intra-rater and inter-rater reliability.
Hyperemia score correlation with UC disease activity | 1 day
  Hyperemia on Doppler EUS to assess inflammatory changes in UC patients with active inflammation compared to quiescent disease

CONTACTS AND LOCATIONS:
Overall Officials: Brian Yan, MD, Principal Investigator — Western University
Locations (1):
- St. Joseph's Health Care, London, Ontario, Canada

REFERENCES:
- [Background] Parente F, Molteni M, Marino B, Colli A, Ardizzone S, Greco S, Sampietro G, Foschi D, Gallus S. Are colonoscopy and bowel ultrasound useful for assessing response to short-term therapy and predicting disease outcome of moderate-to-severe forms of ulcerative colitis?: a prospective study. Am J Gastroenterol. 2010 May;105(5):1150-7. doi: 10.1038/ajg.2009.672. Epub 2009 Dec 8. PMID 19997096
- [Background] Tsuga K, Haruma K, Fujimura J, Hata J, Tani H, Tanaka S, Sumii K, Kajiyama G. Evaluation of the colorectal wall in normal subjects and patients with ulcerative colitis using an ultrasonic catheter probe. Gastrointest Endosc. 1998 Nov;48(5):477-84. doi: 10.1016/s0016-5107(98)70088-4. PMID 9831835
- [Background] Higaki S, Nohara H, Saitoh Y, Akazawa A, Yanai H, Yoshida T, Okita K. Increased rectal wall thickness may predict relapse in ulcerative colitis: a pilot follow-up study by ultrasonographic colonoscopy. Endoscopy. 2002 Mar;34(3):212-9. doi: 10.1055/s-2002-20293. PMID 11870572
- [Background] Yoshizawa S, Kobayashi K, Katsumata T, Saigenji K, Okayasu I. Clinical usefulness of EUS for active ulcerative colitis. Gastrointest Endosc. 2007 Feb;65(2):253-60. doi: 10.1016/j.gie.2005.10.037. PMID 17258984
- [Background] Hurlstone DP, Sanders DS, Lobo AJ, McAlindon ME, Cross SS. Prospective evaluation of high-frequency mini-probe ultrasound colonoscopic imaging in ulcerative colitis: a valid tool for predicting clinical severity. Eur J Gastroenterol Hepatol. 2005 Dec;17(12):1325-31. doi: 10.1097/00042737-200512000-00010. PMID 16292085
- [Background] D'Haens G, Sandborn WJ, Feagan BG, Geboes K, Hanauer SB, Irvine EJ, Lemann M, Marteau P, Rutgeerts P, Scholmerich J, Sutherland LR. A review of activity indices and efficacy end points for clinical trials of medical therapy in adults with ulcerative colitis. Gastroenterology. 2007 Feb;132(2):763-86. doi: 10.1053/j.gastro.2006.12.038. Epub 2006 Dec 20. No abstract available. PMID 17258735
- [Background] Travis SP, Schnell D, Krzeski P, Abreu MT, Altman DG, Colombel JF, Feagan BG, Hanauer SB, Lemann M, Lichtenstein GR, Marteau PR, Reinisch W, Sands BE, Yacyshyn BR, Bernhardt CA, Mary JY, Sandborn WJ. Developing an instrument to assess the endoscopic severity of ulcerative colitis: the Ulcerative Colitis Endoscopic Index of Severity (UCEIS). Gut. 2012 Apr;61(4):535-42. doi: 10.1136/gutjnl-2011-300486. Epub 2011 Oct 13. PMID 21997563
- [Background] Geboes K, Riddell R, Ost A, Jensfelt B, Persson T, Lofberg R. A reproducible grading scale for histological assessment of inflammation in ulcerative colitis. Gut. 2000 Sep;47(3):404-9. doi: 10.1136/gut.47.3.404. PMID 10940279
- [Background] Kornbluth A, Sachar DB; Practice Parameters Committee of the American College of Gastroenterology. Ulcerative colitis practice guidelines in adults (update): American College of Gastroenterology, Practice Parameters Committee. Am J Gastroenterol. 2004 Jul;99(7):1371-85. doi: 10.1111/j.1572-0241.2004.40036.x. PMID 15233681
- [Background] Lichtenstein GR, Abreu MT, Cohen R, Tremaine W; American Gastroenterological Association. American Gastroenterological Association Institute technical review on corticosteroids, immunomodulators, and infliximab in inflammatory bowel disease. Gastroenterology. 2006 Mar;130(3):940-87. doi: 10.1053/j.gastro.2006.01.048. No abstract available. PMID 16530532
- [Background] Langhorst J, Elsenbruch S, Koelzer J, Rueffer A, Michalsen A, Dobos GJ. Noninvasive markers in the assessment of intestinal inflammation in inflammatory bowel diseases: performance of fecal lactoferrin, calprotectin, and PMN-elastase, CRP, and clinical indices. Am J Gastroenterol. 2008 Jan;103(1):162-9. doi: 10.1111/j.1572-0241.2007.01556.x. Epub 2007 Oct 4. PMID 17916108
- [Derived] Yan B, Feagan B, Teriaky A, Mosli M, Mohamed R, Williams G, Yeung E, Yong E, Haig A, Sey M, Stitt L, Zou GY, Jairath V. Reliability of EUS indices to detect inflammation in ulcerative colitis. Gastrointest Endosc. 2017 Dec;86(6):1079-1087. doi: 10.1016/j.gie.2017.07.035. Epub 2017 Jul 29. PMID 28760533